CLINICAL TRIAL: NCT02779777
Title: An Adaptive Phase 2 Study of Tipifarnib in Subjects With Myelodysplastic Syndromes
Brief Title: Tipifarnib in Subjects With Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Kura Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KO-TIP-003
Record Dates: First submitted 2016-05-10; First posted 2016-05-20 (Estimated); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — tipifarnib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regimen 1: Tipifarnib (Experimental): 600 mg twice daily (bid) for 7 days on Days 1-7 in 28 day cycles.
  Interventions: Drug: Tipifarnib
- Regimen 2: Tipifarnib (Experimental): 300 mg bid for 21 days on Days 1-21 in 28 day cycles.
  Interventions: Drug: Tipifarnib

INTERVENTIONS:
Drug: Tipifarnib — Oral tablet
  Other Names: Zarnesta

SUMMARY:
This is a Phase 2 randomized, open-label, two-stage study designed to investigate the antitumor activity of tipifarnib in approximately 36 eligible subjects with MDS who have no known curative treatment. Subjects will be randomized to receive tipifarnib orally with food according to one of 2 treatment regimens.

DETAILED DESCRIPTION:
This Phase 2 study will investigate the antitumor activity in terms of ORR of tipifarnib in approximately 36 eligible subjects with MDS who have no known curative treatment. Eligible subjects may have received no more than 2 prior systemic regimens. Subjects will be randomized to receive tipifarnib orally with food according to one of 2 dose regimens. In the absence of unmanageable toxicities, subjects may continue to receive tipifarnib treatment until disease progression.

Disease assessments will be performed at screening and at least once every approximately 12 weeks starting at the end of cycle 3. Determination of ORR will be assessed by the Investigator according to the MDS International Working Group (IWG) criteria (Cheson 2006). Upon disease progression, all subjects in the study will be followed approximately every 12 weeks for survival and the use of subsequent therapy until either death or 12 months after accrual of the study has been completed, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age.
* Documented pathological evidence of MDS as defined by the World Health Organization (WHO) criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* Subjects have no known curative treatment.
* Subject is willing and able to comply with scheduled visits, treatment plans, laboratory tests and other procedures (including bone marrow assessments).
* At least 1 week since the last systemic therapy regimen prior to Cycle 1 Day 1. Subjects must have recovered to NCI CTCAE v. 4.03 < Grade 2 from all acute toxicities (excluding Grade 2 toxicities that are not considered a safety risk by the Sponsor and Investigator) or toxicity must be deemed irreversible by the Investigator.
* Acceptable hematological function:

  1. Absolute neutrophil count < 1000/mm3
  2. Platelet count > 20,000/mm3
* Acceptable liver function:

  1. Total or direct bilirubin ≤ 1.5 times upper limit of normal (x ULN); does not apply to subjects with Gilbert's syndrome diagnosed as per institutional guidelines.
  2. AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN.
* Acceptable renal function with serum creatinine ≤ 1.5 x ULN or a calculated creatinine clearance ≥ 60 mL/min using the Cockcroft-Gault or Modification of Diet in Renal Disease formulas.
* Female subjects must be:

  1. Of non-child-bearing potential (surgically sterilized or at least 2 years post-menopausal); or
  2. If of child-bearing potential, subject must use a highly effective method of contraception, such as combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner or sexual abstinence. Both females and male subjects with female partners of child-bearing potential must agree to use a highly effective method of contraception for 2 weeks prior to screening, during, and at least 4 weeks after last dose of trial medication. Female subjects must have a negative serum or urine pregnancy test within 72 hours prior to start of trial medication.
  3. Not breast feeding at any time during the study.
* Written and voluntary informed consent understood, signed and dated.

Exclusion Criteria:

* Known prior progression to acute myeloid leukemia (AML), defined by at least 20% blasts in the blood or bone marrow.
* Myelodysplastic or myeloproliferative syndrome other than MDS.
* More than two prior systemic regimens for MDS. Prior systemic regimens are those that are considered standard of care for the treatment of MDS, have been received at standard doses for at least one full treatment cycle and exclude ESA.
* Prior cytoreductive therapy for blast reduction.
* Participation in any interventional study within 1 week or 5 half lives (whichever is longer) of Cycle 1 Day 1.
* Ongoing treatment with an anticancer agent for MDS not contemplated in this protocol.
* Prior treatment (at least 1 full treatment cycle) with a farnesyltransferase inhibitor.
* Clinically significant anemia due to iron, B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or gastrointestinal bleeding. If marrow stain for iron is not available, the transferrin saturation (iron/total iron binding capacity Fe/TIBC) must be >20% or serum ferritin must be >100 ng/dL.
* Active coronary artery disease requiring treatment, myocardial infarction within the prior year, New York Heart Association grade III or greater congestive heart failure, cerebro-vascular attack within the prior year, or current serious cardiac arrhythmia requiring medication except atrial fibrillation.
* Major surgery, other than diagnostic surgery, within 2 weeks prior to Cycle 1 Day 1, without complete recovery.
* Active, concurrent malignancy requiring radiation, chemotherapy, or immunotherapy (excluding non-melanoma skin cancer, adjuvant hormonal therapy for breast cancer and hormonal treatment for castration sensitive prostate cancer).
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy. Known infection with human immunodeficiency virus (HIV), or an active infection with hepatitis B or hepatitis C.
* Subjects who have exhibited allergic reactions to tipifarnib, or structural compounds similar to tipifarnib or to its excipients.
* Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study.
* The subject has legal incapacity or limited legal capacity.
* Significantly altered mental status that would limit the understanding or rendering of informed consent and compliance with the requirements of this protocol. Unwillingness or inability to comply with the study protocol for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects affected by myelodysplastic syndromes (MDS) were recruited across 2 sites in the United States between June 2016 and August 2018.
Pre-assignment Details: This study included a screening period, treatment period (28-day cycles until disease progression), end of treatment visit, follow-up visit (for subjects who terminated treatment for reasons other than death or disease progression), and follow-up contact (upon disease progression, all subjects were followed approximately every 12 weeks for survival and use of subsequent therapy until either death or accrual in the subject's study cohort was completed, whichever occurred first).
Groups:
- Original Cohort: Subjects prior to Amendment 3 were considered to be the Original Cohort. Prior to Amendment 3 this was a non-randomized study with 900 twice daily (BID) (Days 1-7 and 15-21) in 28 day cycles, allowing for adjustments in dosing/schedule based on patient tolerability.
- Regimen 2: Tipifarnib: 300 mg BID for 21 days on Days 1-21 in 28 day cycles (ie, 3 weeks on/1 weeks off).
Period: Overall Study
Arm/Group | Original Cohort | Regimen 1: Tipifarnib | Regimen 2: Tipifarnib
Started | 14 | 1 | 1
Completed | 0 | 0 | 0
Not Completed | 14 | 1 | 1
Not completed — Disease Progression | 1 | 0 | 0
Not completed — Adverse Event | 3 | 1 | 0
Not completed — Physician Decision | 9 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Regimen 1: Tipifarnib: 600 mg BID for 7 days on Days 1-7 in 28 day cycles (ie, 1 week on/3 weeks off).
- Regimen 2: Tipifarnib: 300 mg BID for 21 days on Days 1-21 in 28 day cycles (ie, 3 weeks on/1 week off).
- Total: Total of all reporting groups
Arm/Group | Original Cohort | Regimen 1: Tipifarnib | Regimen 2: Tipifarnib | Total
Number analyzed (Participants) | 14 | 1 | 1 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.2 (7.5) | 76.6 (NA) — Only 1 subject was analyzed, therefore standard deviation cannot be determined. | 68.9 (NA) — Only 1 subject was analyzed, therefore standard deviation cannot be determined. | 71.4 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 0 | 6
  Male | 8 | 1 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 13 | 1 | 1 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2
  White | 10 | 1 | 0 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
ECOG Performance Status [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without hesitation.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light housework, office work.
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Participants
    0 | 12 | 1 | 0 | 13
    1 | 1 | 0 | 1 | 2
    2 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was assessed by the investigator and included complete response (CR), partial response (PR), marrow complete remission (MR), and hematologic improvement (HI) according to the MDS International Working Group (IWG) criteria.
Time Frame: 1 year
Population: Full analysis set (FAS) includes subjects enrolled in Protocol Amendment 3 (version 09 Jul 2017) and received at least one dose of tipifarnib.
Measure: Count of Participants; unit: Participants
Groups:
- Original Cohort: Subjects prior to Amendment 3 were considered to be the Original Cohort. Prior to Amendment 3 this was a non-randomized study with 900 BID (Days 1-7 and 15-21) in 28 day cycles, allowing for adjustments in dosing/schedule based on patient tolerability.
Arm/Group | Original Cohort | Regimen 1: Tipifarnib | Regimen 2: Tipifarnib
Number analyzed (Participants) | 0 | 1 | 1
Participants | 0 | 0 | 0

2. Secondary Outcome: Rate of Transfusion Independence
Description: Rate of transfusion independence is defined as number of participants with transfusion independence at any response assessment over 1 year.
Time Frame: 1 year
Population: FAS includes subjects enrolled in Protocol Amendment 3 (version 09 Jul 2017) and received at least one dose of tipifarnib.
Measure: Count of Participants; unit: Participants
Groups:
- Regimen 1: Tipifarnib: 600 mg BID for 7 days on Days 1-7 in 28 day cycles.
Arm/Group | Original Cohort | Regimen 1: Tipifarnib | Regimen 2: Tipifarnib
Number analyzed (Participants) | 0 | 1 | 1
Participants | 0 | 0 | 0

3. Secondary Outcome: Duration of Transfusion Independence
Description: Duration of transfusion independence is defined as the period of time where participants achieved transfusion independence.
Time Frame: 1 year
Population: as for outcome 2
Arm/Group | Original Cohort | Regimen 1: Tipifarnib | Regimen 2: Tipifarnib
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Hematologic Improvement
Description: Number of subjects who experienced hematologic improvements (erythroid response, platelet response, or neutrophil response).
Time Frame: 1 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Original Cohort | Regimen 1: Tipifarnib | Regimen 2: Tipifarnib
Number analyzed (Participants) | 0 | 1 | 1
Participants | 0 | 0 | 1

5. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the number of days from the start date of response (whichever response is achieved first) to the first date that progressive disease is objectively documented.
Time Frame: 1 year
Population: as for outcome 2
Arm/Group | Original Cohort | Regimen 1: Tipifarnib | Regimen 2: Tipifarnib
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Progression-free Survival (PFS) at 1 Year
Description: PFS is defined as the time (in months) from enrollment to either first observation of progressive disease or occurrence of death due to any cause within 1 year (approximately 4 time intervals for disease assessments) of either first administration of tipifarnib or the last disease assessment.
Time Frame: 1 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Original Cohort | Regimen 1: Tipifarnib | Regimen 2: Tipifarnib
Number analyzed (Participants) | 0 | 1 | 1
Participants |  | 0 | 0

7. Secondary Outcome: Overall Survival (OS) at 1 Year
Description: OS is defined as the time (in months) from enrollment to occurrence of death due to any cause within 1 year (approximately 4 time intervals for disease assessments) of either first administration of tipifarnib or the last disease assessment.
Time Frame: 1 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Original Cohort | Regimen 1: Tipifarnib | Regimen 2: Tipifarnib
Number analyzed (Participants) | 0 | 1 | 1
Participants |  | 0 | 0

8. Secondary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs are defined as AEs that started on or after the first dose of study drug and within approximately 30 days of the last administration of study drug. AEs were summarized by the number and percentage of subjects who experienced the event, according to system organ class and preferred term. A subject reporting multiple cases of the same AE will be counted once within each system organ class and similarly counted once within each preferred term.
Time Frame: 1 year
Population: The All Subjects as Treated (ASaT) population consisted of all enrolled subjects who received at least 1 dose of tipifarnib.
Measure: Count of Participants; unit: Participants
Arm/Group | Original Cohort | Regimen 1: Tipifarnib | Regimen 2: Tipifarnib
Number analyzed (Participants) | 14 | 1 | 1
Participants
  Subjects with one or more TEAE | 14 | 1 | 1
  Subjects with one or more study drug-related TEAE | 14 | 1 | 1
  Subjects with one or more serious TEAE | 7 | 0 | 0
  Subjects with one or more study drug-related serious TEAE | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: The ASaT population consisted of all enrolled subjects who received at least 1 dose of tipifarnib.
Arm/Group | Original Cohort | Regimen 1: Tipifarnib | Regimen 2: Tipifarnib
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 7/14 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 14/14 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Original Cohort (N=14) | Regimen 1: Tipifarnib (N=1) | Regimen 2: Tipifarnib (N=1)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Original Cohort (N=14) | Regimen 1: Tipifarnib (N=1) | Regimen 2: Tipifarnib (N=1)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (9) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 6 (6) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (5) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Iron overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are agreements in place between clinical trial sites and the Sponsor (or its agents) that govern discussion or publication of trial results by the sites or their employees after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT02779777/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT02779777/SAP_001.pdf